CLINICAL TRIAL: NCT01675817
Title: Evaluation of Heparin Rebound in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: R-10-190; 16949E (Other: REB)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2012-09

CONDITIONS: Coagulation Delay
Keywords: heparin rebound; protamine; cardiopulmonary bypass; cardiac surgery; anti-Xa; anti-IIa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent work has shown that heparin rebound is common after cardiac surgery.

The exact doze of protamine required to neutralize heparin at the end of CPB is unknown. Besides, the precise doze of protamine to treat heparin rebound is also unknown. It is also unknown if precise titration of protamine perioperatively in cardiac surgery can influence transfusion requirements after cardiac surgery.

DETAILED DESCRIPTION:
This study will assess how much protamine is required to neutralize residual heparin perioperatively in cardiac surgery through measurement of functional assays of heparin (anti-Xa and anti-IIa levels). In the first phase of this study, protamine titration assays will be carried out on normal pooled plasma incubated with heparin in the laboratory.

Once the correct dose of protamine required to neutralize the heparin is established in the laboratory, the second phase will begin. Herein, plasma samples from patients undergoing cardiac surgery (with anticoagulation with two different commercial preparations of heparin) will be evaluated for residual heparin (Anti-Xa and anti-IIa levels). Protamine titration assays wil then be carried out in vitro to assess neutralization of heparin.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Written consent
* Scheduled for cardiac surgery under CPB (cardiopulmonary bypass)--(elective or emergency)
* 10 patients undergoing cardiac surgery where CPB time is anticipated to be short (isolated primary CABG (coronary artery bypass graft);isolated mitral-valve repair or aortic-valve replacement)
* 10 patients undergoing cardiac surgery where CPB time is anticipated to be longer (CABG + valve surgery combined; reoperations)

Exclusion Criteria:

* Known coagulopathies
* Liver dysfunction
* Patients receiving unfractionated or low molecular weight heparin thrombin inhibitors, warfarin, antiplatelets within the past 7 days
* Patients expected to undergo hypothermic CPB or circulatory arrest

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Taneja, MD, FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Dr. Ravi Taneja, London, Ontario, Canada

REFERENCES:
- [Derived] Taneja R, Berry L, Pappu U, Stitt L, Sayal P, Allen P, Hoogendoorn H, Chan A. Protamine requirements in cardiac surgery: effect of changes in the heparin reference standard. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1227-32. doi: 10.1053/j.jvca.2014.04.024. PMID 25281041